CLINICAL TRIAL: NCT01988155
Title: Eccentric Exercise Versus Eccentric Exercise and Astym® in the Management of Insertional Achilles Tendinopathy: A Randomized Controlled Trial
Brief Title: Eccentric Exercise Versus Eccentric Exercise and Astym for Insertional Achilles Tendinopathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University Health Ball Memorial Hospital Rehabiliation Services (Other)
Collaborators: Performance Dynamics Inc (Unknown)
Responsible Party: Principal Investigator, Joshua McCormack, Physical Therapist, Indiana University Health Ball Memorial Hospital Rehabiliation Services
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 13-928
Record Dates: First submitted 2013-11-08; First posted 2013-11-20 (Estimated); Last update posted 2016-02-23 (Estimated); Status verified 2016-02

CONDITIONS: Insertional Achilles Tendinopathy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Eccentric Exericse (Active Comparator)
  Interventions: Other: Eccentric Exercise
- Astym (Experimental)
  Interventions: Other: Astym

INTERVENTIONS:
Other: Eccentric Exercise — Subjects in the eccentric exercise group will be instructed to perform the modified Alfredson eccentric protocol for insertional Achilles tendinopathy. To perform the eccentric exercise, subjects will be instructed to stand upright with one hand on the wall or a chair for support as needed. A heel raise exercise is then performed with the non-painful leg. Once in the elevated position, subjects are instructed to transfer all of their body weight to the painful leg and slowly lower their heel to the floor while keeping their knee extended. The eccentric exercise program will consist of 3 sets of 15 repetitions performed per session. Subjects will perform 2 sessions per day for a total of 12 weeks and a log will be kept to monitor compliance. In order to partially control for the effect of regular contact with a therapist, subjects in the control group will be contacted by telephone one time per week to discuss their progress with the program and address any questions they may have.
  Arms: Eccentric Exericse
Other: Astym — In addition to performing the same eccentric protocol as the eccentric exercise group, subjects in the Astym group will also be seen in the clinic two times per week. Astym treatment will be performed per the foot, ankle, and knee protocol as described in the Astym clinical manual. During the first visit each week, the eccentric exercise protocol will be orally reviewed to match the one time per week phone education received by the eccentric only group. Astym treatment will continue for up to six weeks but may be discontinued early if a subject scores 90 or above on the VISA-A. Subjects in the Astym group will be required to continue with the eccentric exercise protocol for the full 12 weeks even in Astym is discontinued early.
  Arms: Astym

SUMMARY:
The purpose of this research study is to determine if Astym® treatment is an effective treatment for patients with Achilles pain. The usual treatment for this condition is a specific exercise program that has been previously shown to be effective. The research team is trying to determine if combining Astym with the exercise program is more effective than exercise program only.

The main hypothesis for this study is that Astym plus eccentric exercise will be more effective than eccentric exercise alone at improving pain and function in patients with insertional Achilles tendinopathy.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of insertional AT as a primary complaint*
* symptom duration of at least 6 weeks
* VISA-A score of 78 or lower

  * he presence of insertional AT will be clinically determined by the primary investigator using the following criteria: pain at or within 2 cm of the posterior calcaneal insertion of the Achilles tendon along with localized tenderness and a subjective report of decreased activity levels secondary to Achilles pain.

Exclusion Criteria:

* prior treatment with eccentric exercise or Astym for Achilles tendinopathy
* currently taking anticoagulant medication
* usage of fluoroquinolone antibiotics in the previous six months
* previous Achilles surgery on the involved side
* bilateral symptoms
* pregnancy
* worker's compensation or liability cases
* peripheral neuropathy
* signs of lumbar radiculopathy
* inability to complete the required outcomes forms or comply with the recommended treatment regimen

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2013-12; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Victorian Institute of Sport Assessment- Achilles Specific Questionnaire (VISA-A) | 12 weeks

SECONDARY OUTCOMES:
Numeric Pain Rating Scale (NPRS) | 12 weeks
  Average of Best, Worst, and Current pain from 0-10
Global Rating of Change Score (GROC) | 12 weeks

OTHER OUTCOMES:
Percent Recovered | 12 weeks
  The percentage of subjects in each group that reach 90 or higher on the VISA-A by 12 weeks.
Percent Improved | 12 weeks
  The percentage of subjects in each group that improve by the MCID (12 points) or more on the VISA-A at 12 weeks.
Victorian Institute of Sport Assessment- Achilles Specific Questionnaire (VISA-A) | 4 weeks
Victorian Institute of Sport Assessment- Achilles Specific Questionnaire (VISA-A) | 8 weeks
Victorian Institute of Sport Assessment- Achilles Specific Questionnaire (VISA-A) | 26 weeks
Victorian Institute of Sport Assessment- Achilles Specific Questionnaire (VISA-A) | 52 weeks
Numeric Pain Rating Scale (NPRS) | 4 weeks
  Average of Best, Worst, and Current pain from 0-10
Numeric Pain Rating Scale (NPRS) | 26 weeks
  Average of Best, Worst, and Current pain from 0-10
Numeric Pain Rating Scale (NPRS) | 52 weeks
  Average of Best, Worst, and Current pain from 0-10
Numeric Pain Rating Scale (NPRS) | 8 weeks
  Average of Best, Worst, and Current pain from 0-10

CONTACTS AND LOCATIONS:
Locations (1):
- IU Health BMH Rehab at CIO, Muncie, Indiana, United States